CLINICAL TRIAL: NCT06744621
Title: Glucose Monitoring for A1GDM
Brief Title: Glucose Frequent of A1GDM in Labor
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Thomas Owens, Maternal Fetal Medicine Fellow, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-24-01116
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Gestational Diabetes, Controlled by Diet
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Infrequent: Patients will undergo one fingerstick on admission for their labor process.
  Interventions: Other: Fingerstick
- Frequent: Patients will undergo fingersticks every 4 hours in latent labor and 2 hour in active labor during their labor process.
  Interventions: Other: Fingerstick

INTERVENTIONS:
Other: Fingerstick — fingersticks during their labor process

SUMMARY:
This is a prospective double arm study in patients with Gestational Diabetes Mellitus (GDM) utilizing frequent (single fingerstick on admission) vs infrequent glucose monitoring in labor (q 4 hours in latent labor and every 2 hours in active labor). Primary Objective: The primary outcome is glucose value of the neonate at birth. Secondary Objectives: Determine rates of insulin requirements within different monitoring techniques. Determine if there is a difference in neonatal intensive care unit (NICU) admission within different monitoring techniques. Determine neonatal blood glucose concentrations at 24 hours of life, number of glucose treatments, and neonatal hyperbilirubinemia. Secondary characteristics to be viewed for each diagnosis; BMI, race, age, and parity.

ELIGIBILITY:
Inclusion Criteria:

* All female patients of reproductive age (menarche-menopause: 18-51 years) who have the diagnosis diet controlled GDM
* Patient with singleton gestation presenting in labor or for induction
* Patients who had "good" glucose control and were A1GDM. Good Control;

  * - Patient with overall outpatient glucose average of less than 100
  * - No evidence of fetopathy, large for gestational age or polyhydramnios.
  * - Hgb A1c <5.7

Exclusion Criteria:

• If patient's admission accu check is >120

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient with A1GDM (diet controlled gestational diabetes)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Neonatal glucose level | at 24 hours

SECONDARY OUTCOMES:
Number of neonates requiring insulin | at 24 hours
Number of NICU admissions | at 24 hours
Number of glucose treatments | at 24 hours
Number of neonatal with hyperbilirubinemia | at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Owens, MD, Principal Investigator — Mount Sinai West
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No